CLINICAL TRIAL: NCT00398788
Title: An Open-Label, Repeated-Dose Trial to Characterize the Efficacy and Safety, and Impact on Quality of Life Measures of Dilaudid CR (Hydromorphone HCI) in Patients With Chronic Low Back Pain
Brief Title: A Study on Efficacy (Effectiveness), Safety, and Impact on Quality of Life Measures of Dilaudid CR (Controlled Release);, Hydromorphone HCl in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013255
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Low Back Pain
Keywords: Pain
MeSH Terms: conditions — Low Back Pain; Pain

INTERVENTIONS:
Drug: OROS® hydromorphone HCL; Dilaudid CR (controlled release); Dilaudid IR (immediate release) as rescue medicine

SUMMARY:
The purpose of the study was to characterize the safety, effectiveness, and impact on quality of life (QOL) measures of OROSÂ® hydromorphone HCL in patients with chronic low back pain.

DETAILED DESCRIPTION:
This study was a short-term, non-randomized (each patient was assigned the same treatment from phase I through phase III by the researchers), non-comparative, open-label, repeated dose study of OROS® hydromorphone HCL consisting of 3 phases: Phase 1 - prior opioid stabilization phase (2-7 days); Phase 2 - OROS® hydromorphone HCL conversion, titration, and stabilization phase (3 - 14 days); Phase 3 - OROS® hydromorphone HCL maintenance therapy phase (28 days) Before Phase 1, patients must have had no change in their prescribed opioid regimen over the prior 30 days. During Phase 1, patients were to have demonstrated 2 consecutive days of stable baseline oral or transdermal opioid medication.

During Phase 2, patients requiring =96 mg OROS® hydromorphone HCL every 24 hours converted to a once-daily dosing OROS® hydromorphone HCL dose at approximately a 5:1 morphine to hydromorphone equivalent ratio. OROS® hydromorphone HCL dose titration (25-100% baseline dose) was allowed every 2 days to achieve stabilization. OROS® hydromorphone HCL dose reduction was allowed during Phases 2 and 3 for opioid-related adverse events (AEs). Rescue medication, Dilaudid IR (immediate release) was allowed during all 3 phases. During Phase 3, patients attended 4 weekly study visits to provide diary information about study medication and rescue medication usage, daily pain relief scores and adverse events, and to receive weekly supplies of study medications. OROS® hydromorphone HCL tablets of 8,16, 32, or 64 mg depending on Phase I stable baseline oral or transdermal opioid medication, 2-7 days; study drug dose titration was allowed every 2 days to achieve stabilization in Phase II, 3-14 days; Phase III , maintenance therapy phase 28 days; study drug dose reduction was allowed during Phase 2 and 3 for opioid-related adverse events. Rescue medication of Dilaudid IR (immediate release) 2, 4, 8mg tablets were allowed during all phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic low back pain who were currently receiving strong oral or transdermal opioid analgesics on a daily basis, or patients suitable for advancement of therapy to step 3 of the World Health Organization (WHO) analgesic ladder were considered for enrollment in the study. Patients requiring >8 and =96 mg of OROS® hydromorphone HCL every 24 hours were enrolled in the study.

Exclusion Criteria:

* Patients intolerant or hypersensitive to hydromorphone or other opioid agonists and patients with a known history of alcohol or drug abuse within the previous year were excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
The mean pain relief rating derived from daily recorded patient diaries during the 4 week maintenance phase;

SECONDARY OUTCOMES:
The overall global evaluation and Brief Pain Inventory (BPI) of study drug, as assessed by both patients and Investigators at weekly visits during the 4 week maintenance phase.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Wallace M, Skowronski R, Khanna S, Tudor IC, Thipphawong J. Efficacy and safety evaluation of once-daily OROS hydromorphone in patients with chronic low back pain: a pilot open-label study (DO-127). Curr Med Res Opin. 2007 May;23(5):981-9. doi: 10.1185/030079907x182040. PMID 17519065